CLINICAL TRIAL: NCT07392138
Title: Understanding Newborn-Mother Synchrony at Home: Feasibility of Remote Monitoring
Status: Not yet recruiting | Type: Observational
Sponsor: University of Turku (Other)
Responsible Party: Principal Investigator, Anna Axelin, Professor, University of Turku
Other Study IDs: #476745
Record Dates: First submitted 2026-01-12; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Synchrony

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Newborn
  Interventions: Other: Using monitoring devices
- Mother
  Interventions: Other: Using monitoring devices

INTERVENTIONS:
Other: Using monitoring devices — During the data collection, mother and newborn are using the monitoring devices listed in study description.

SUMMARY:
Parents and newborns influence each other in a dynamic interaction that can be described as synchrony. Synchrony between a newborn and mother refers to the dynamic and reciprocal adaptation between the newborn and mother. In this synchrony, the mother is highly receptive and sensitive to the newborn's signals, feelings, and needs. The aim of this study is to investigate the physiological and behavioral synchrony between newborns and their mothers, and to investigate the connection between maternal heart rate variability and postpartum depression symptoms in the home environment and to evaluate the suitability of remote monitoring devices for use in the home environment.

The study participants consist of 30 newborns and 30 mothers. The inclusion criteria for newborns are: 1) informed consent from the newborn's parents/guardians 2) the newborn's health status has been confirmed as normal during hospital monitoring, and 3) the newborn is less than one month old. The inclusion criteria for mothers are: 1) ability to participate in Finnish, and 2) the mother has access to an Android smartphone.

Data collection will be carried out using the following remote monitoring methods: Emfit smart mattress, Zoundream Cry analyses technology, Polar Verity Sense sensor, and Empatica EmbracePlus sensor. In addition, data will be collected using background information forms, a maternal stress scale (PSS-4), a diary completed by the mother, a maternal depression questionnaire (EPDS), and questionnaires measuring the suitability of remote monitoring in the home environment, and a thematic interview. In addition, at the end of the data collection phase, the mothers participating in the study will try out the Companion App, which displays sample data on the well-being of newborns, and respond to a questionnaire on the usability of the app.

ELIGIBILITY:
Inclusion Criteria, mothers:

* ability to participate in Finnish
* Android smart phone available

Inclusion Criteria, newborns:

* received informed consent from both parents/guardians
* the newborn's health has been stated normal during hospital stay
* the newborn is < 1-month of age

Exclusion Criteria, both (mother and newborn):

Not meeting the inclusion criteria

Min Age: 0 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Study population consists of mother-newborn pairs.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Physiological synchrony | 24 hours
  Measuring correlation between mother heart rate (mHR (unit: BPM)) and heart rate variability (mHRV (unit ms)) and newborn heart rate (bHR (unit: BPM)) and heart rate variability (bHRV (unit: ms)).

SECONDARY OUTCOMES:
Behavioral synchrony | 24 hours
  Measuring the correlation between mother total sleep duration and duration of different sleep stages and newborn total sleep duration and duration of sleep stages (unit: hours and minutes).
Correlation between mother heart rate variability and depressive symptoms | Duration of data collection varies from 1 to 4 weeks depending on the mother's decision.
  Measuring the correlation between mother heart rate variability (mHRV (units: ms)) and depressive symptoms (points from EPDS scale).
Correlation between mother sleep and depressive symptoms. | Duration of data collection varies from 1 to 4 weeks, depending on the mother's decision.
  Measuring the correlation between the duration of mother sleep stages (unit: hours and minutes) and depressive symptoms (points from EPDS scale).

CONTACTS AND LOCATIONS:
Locations (1):
- Turku University Hospital, Turku, Finland

IPD SHARING:
Plan to Share IPD: No